CLINICAL TRIAL: NCT06821048
Title: A Phase I Clinical Study of Anti-CEA CAR-T (PTC13) Therapy in the Treatment of CEA-positive Advanced Malignant Solid Tumors
Brief Title: Study of CEA Targeting CAR-T (PTC13) in the Treatment of CEA-Positive Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weijia Fang, MD (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Weijia Fang, MD, Principal Investigator, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBC039V1.4
Record Dates: First submitted 2025-02-04; First posted 2025-02-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Stomach Cancer; Pancreatic Cancer; Metastatic Cancer
Keywords: FAST CAR-T; CEA-positive advanced malignant solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraperitoneal infusion of FAST CEA-targeted CAR-T (PTC13) (Experimental): Intraperitoneal infusion of FAST CEA-targeted CAR-T cells (PTC13) by 4 dose levels
  Interventions: Biological: Intraperitoneal infusion of FAST CEA-targeted CAR-T

INTERVENTIONS:
Biological: Intraperitoneal infusion of FAST CEA-targeted CAR-T — Intraperitoneal infusion of FAST CEA-targeted CAR-T (PTC13); Subjects will be treated with Fludarabine and Cyclophosphamide based lymphodepleting chemotherapy before CAR-T cell infusion.

SUMMARY:
This is a phase I clinical study to evaluate the safety and tolerability of FAST targeted chimeric antigen receptor (CAR)-T cells (PTC13) in patients with carcinoembryonic antigen (CEA)-positive advanced malignant solid tumors, and to obtain the maximum tolerated dose of FAST CAR-T (PTC13) and phase II Recommended dose.

DETAILED DESCRIPTION:
This is a single-center, open-label, dose-escalation and expansion study. The study includes one intraperitoneal infusion group only, with four dose levels: 2.0×10⁵ CAR+ cells/kg, 3.0×10⁵ CAR+ cells/kg, 4.0×10⁵ CAR+ cells/kg, and 5.0×10⁵ CAR+ cells/kg. Each dose level will initially enroll 3 to 6 patients using a standard 3+3 design to preliminarily evaluate safety and efficacy. Based on the comprehensive assessment by investigators and the technical collaborators, 1 to 2 recommended dose levels will be selected for dose expansion. In the expansion phase, an additional 6 to 12 patients will be enrolled to further evaluate safety and efficacy. The total planned enrollment is approximately 18 to 36 patients. Priority will be given to patients with peritoneal metastases from colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for the study:

1. Age≥18 years, regardless of gender.
2. Diagnosed with advanced, metastatic, or recurrent malignant tumors confirmed by histology or pathology, primarily including colorectal cancer, esophageal cancer, gastric cancer, pancreatic cancer, lung cancer, or cholangiocarcinoma.
3. Failure of at least second-line standard therapy (due to disease progression or intolerance, such as surgery, chemotherapy, radiotherapy, etc.) or a lack of effective treatment options.
4. Immunohistochemical staining of tumor samples within 3 months confirming CEA positivity (distinct membrane staining with a positivity rate of≥10%); if the immunohistochemical result of the tumor sample is more than 3 months old at the time of screening (distinct membrane staining with a positivity rate of≥10%), the patient's serum CEA must exceed 10µg/L.
5. At least one evaluable lesion according to RECIST 1.1 criteria.
6. ECOG score of 0-2 (Appendix 2).
7. No severe psychiatric disorders.
8. Unless specifically stated otherwise, subjects' major organ functions must meet the following conditions:

   1. Blood routine: WBC>2.0×109/L, neutrophils>0.8×109/L, lymphocytes>0.5×109/L, platelets>50×109/L, hemoglobin>90g/L;
   2. Cardiac function: Echocardiography indicating a left ventricular ejection fraction≥50%, and no significant abnormalities on electrocardiogram;
   3. Renal function: Serum creatinine≤2.0×ULN;
   4. Liver function: ALT and AST ≤3.0×ULN (may be relaxed to≤5.0×ULN if liver tumor infiltration is present);
   5. Total bilirubin≤2.0×ULN;
   6. Oxygen saturation>92% without supplemental oxygen. 9. Eligible for apheresis or venous blood collection, with no contraindications for cell collection.

      10. Subjects agree to use reliable and effective contraceptive methods from signing the informed consent form until 1 year after receiving CAR-T cell infusion (excluding natural family planning methods).

      11. The patient or their guardian agree to participate in this clinical trial and signs the ICF, indicating an understanding of the trial's purpose and procedures and willingness to participate.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Clinically symptomatic central nervous system or leptomeningeal metastasis at the time of screening, or other evidence suggesting that central nervous system or leptomeningeal metastases are not controlled, as judged unsuitable for inclusion by the investigator.
2. Participation in another clinical study within 1 month prior to screening.
3. Receipt of live attenuated vaccines within 4 weeks prior to screening.
4. Receipt of the following anti-tumor treatments before screening: Chemotherapy, targeted therapy, or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter).
5. Presence of active or uncontrolled infections requiring systemic treatment.
6. Patients with intestinal obstruction, active gastrointestinal bleeding, a history of major gastrointestinal bleeding within 3 months, severe gastroduodenal ulcers, or severe gastrointestinal inflammation such as ulcerative colitis.
7. Toxicity from previous anti-tumor therapy that has not improved to baseline levels or≤Grade 1, except for alopecia or peripheral neuropathy.
8. Presence of any of the following cardiac conditions:

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. Myocardial infarction or coronary artery bypass graft (CABG) within 6 months prior to enrollment;
   3. Clinically significant ventricular arrhythmia or history of unexplained syncope (excluding vasovagal or dehydration-related causes);
   4. History of severe non-ischemic cardiomyopathy.
9. Presence of active autoimmune diseases or other conditions requiring long-term immunosuppressive therapy.
10. Diagnosis of another untreated malignancy within the past 3 years, except for in situ cervical cancer or basal cell carcinoma of the skin.
11. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood hepatitis B virus (HBV) DNA levels exceeding the normal range; positive for hepatitis C virus (HCV) antibodies with peripheral blood HCV RNA levels exceeding the normal range; positive for human immunodeficiency virus (HIV) antibodies; or positive syphilis test.
12. Pregnant or breastfeeding women.
13. Any other conditions deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after CEA-CAR-T cells infusion | 28 days
  Incidence and proportion of adverse events during the trial (evaluated per Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE 5.0) and ASTCT criteria)
Obtain the maximum tolerated dose of CEA-CAR-T cells | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Disease control rate of CAR-T cell preparations in CEA-positive advanced malignancies | 3 months
  including complete response (CR), partial response (PR) and stable disease (SD)
Changes in serum tumor markers of CAR-T cell preparations in CEA-positive advanced malignancies | 3 months
  Tumor markers including CEA、 CA199、 CA125
Pharmacokinetic of CAR-T cells (Cmax) | 1 year
  The highest concentration of CAR-T cells in peripheral blood post-administration.
Pharmacokinetic of CAR-T cells (Tmax) | 1 year
  The time to reach the highest concentration
Pharmacokinetic of CAR-T cells (AUC28d/90d) | 1 year
  Area under the curve at 28 days/90 days
Pharmacodynamic of CAR-T cells | 1 year
  Levels of free CEA in peripheral blood at various time points.

OTHER OUTCOMES:
Objective response rate (ORR) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  Objective response rate includes：CR、PR
Duration of Response (DOR) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  DOR will be assessed from the first assessment of CR/PR/SD to the first assessment of recurrence or progression of the disease or death from any cause
Progress-free survival(PFS) of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression.
Overall survival(OS)of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause
Proportion of tumor cells in tumor tissue of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  The rate of tumor cell in tumor tissue will be measured by biopsy and immunohistochemistry
CEA expression level of CEA- CAR-T treatment in patients with CEA-positive advanced malignancies | 1 year
  The CEA expression in tumor tissue will be measured by biopsy and immunohistochemistry
Changes in the number of tumor-infiltrating immune cells of CEA- CAR-T treatment in patients with CEA-positive | 1 year
  the number of tumor-infiltrating immune cells will be measured by biopsy and immunohistochemistry
Exploration of VOCs in Exhaled Breath After CAR-T Infusion and Their Correlation With Immune-Metabolic Changes | 28 days
  This exploratory study aims to investigate the correlation between volatile organic compounds (VOCs) in exhaled breath and immune-metabolic microenvironment changes following CAR-T cell infusion. Breath samples will be collected at baseline (pre-infusion), and at 0.5h, 1h, 2h, 24h, 7d, 14d (or discharge), and 28d post-infusion. VOCs, including reactive aldehydes (e.g., decanal), ketones, fatty acids, and hydrocarbon gases, will be analyzed using GC-MS and thermal desorption techniques. Biomarkers will be profiled and correlated with immunological and metabolic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, Zhejiang University School of Medicine (FAHZU), Hangzhou, Zhejiang, China